CLINICAL TRIAL: NCT03874572
Title: A Phase I Open Label Study Evaluating the Safety and Feasibility of Allogeneic Mesenchymal Stem Cells for Radiation-induced Hyposalivation and Xerostomia in Previous Oropharynx Cancer Patients
Brief Title: Allogeneic Mesenchymal Stem Cells for Radiation-induced Hyposalivation and Xerostomia/Dry Mouth
Acronym: MESRIX-SAFETY
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Charlotte Lynggaard, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVB2018-2; 2018-003856-19 (EudraCT Number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-09

CONDITIONS: Xerostomia Due to Radiotherapy; Hyposalivation; Xerostomia; Oropharynx Cancer; Salivary Gland Diseases; Dry Mouth; Mesenchymal Stem Cells; Mesenchymal Stromal Cells; Stem Cells
Keywords: Xerostomia Due to Radiotherapy
MeSH Terms: conditions — Xerostomia; Oropharyngeal Neoplasms; Salivary Gland Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic mesenchymal stem/stromal cell therapy (Experimental): Treatment with intra-glandular Injections of allogeneic adipose derived stem cells
  Interventions: Biological: Allogeneic adipose derived stem/stromal cells

INTERVENTIONS:
Biological: Allogeneic adipose derived stem/stromal cells — Culture expanded allogeneic adipose derived stem/stromal cells

SUMMARY:
An investigator-initiated, non-randomized, open label study to investigate the safety, feasibility and tolerability of intraglandular injection of allogeneic mesenchymal stem/stromal cells (MSCs) into the submandibular and parotid glands of the patients with radiation-induced hyposalivation and xerostomia after radiation for a oropharyngeal squamous cell carcinoma

DETAILED DESCRIPTION:
Patients with previous oropharyngeal cancer and radiation-induced hyposalivation and xerostomia (dry mouth syndrome) will receive intraglandular injections of allogeneic adipose-derived MSCs into the submandibular and parotid glands. The trial will be Good Clinical Practice (GCP) Monitored. From healthy donors, MSCs will be produced at a Good Manufacturing Practice (GMP) Facility.

The patients will be followed for four months for safety, tolerability, and efficacy registration. Changes in quality of life, unstimulated, and stimulated whole saliva flow rate, salivary gland function will be assessed. Immune response towards receiving allogeneic MSCs will be evaluated in plasma and saliva. Changes in the composition and quality of the whole saliva will be investigated.

Saliva from the participants will altså be compared to saliva from ten healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years
2. Previous radiotherapy +/- chemotherapy for OPSCC stage I- II (UICC-8, 2017)
3. 2 years' follow-up without recurrence
4. Clinically reduced salivation and hyposalivation, evaluated by a screening
5. Unstimulated salivary flow rate between 0.2mL/min and 0.05mL/min
6. Grade 2-3 xerostomia (CTCAEv5.0)
7. WHO Performance status (PS) 0-1
8. Informed consent

Exclusion Criteria:

1. Any cancer in the previous 4 years (not including OPSCC and basocellular carcinomas)
2. Xerogenic medications
3. Penicillin or Streptomycin allergy
4. Any other diseases of the salivary glands, e.g. Sjögren's syndrome or sialolithiasis
5. Previous parotid or submandibular gland surgery
6. Previous treatment with any type of stem cells
7. Breastfeeding, Pregnancy or planned pregnancy within the next 2 years
8. Smoking within the previous 6 months.
9. Alcohol abuse (consumption must not exceed 7 units/week for women and 14 units/week for men (Danish National board health alcohol guidelines3)
10. Any other disease/condition judged by the investigator to be grounds for exclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of patients with serious adverse events | 4 months
  Registration of number of patients with serious adverse events in a 4 months follow-up period

SECONDARY OUTCOMES:
Immune reponse :Development of donor specific antibodies | 4 months
  Registration of development of tissue antibodies towards donor cells
Efficacy: Change in Unstimulated Whole Salivary flow rate | 4 months
  Unstimulated whole saliva flow rate is assessed by sialometry
Efficacy: Change in Stimulated Whole Salivary flow rate | 4 months
  Unstimulated whole saliva flow rate is assessed by sialometry
Efficacy: Change in quality of life | 4 months
  Change in quality of life evaluted by QLQ-H&N-35 and XQ questionnaires
Efficacy: Salivary gland function | 4 months
  Assessed by salivary gland 99mTc scintigraphy
Efficacy: Change in Saliva composition | 4 months
  Change in inorganic saliva composition
Efficacy: Change in Saliva Proteomics | 4 months
  Change in Saliva proteomics
Efficacy: Change in RNA in Saliva | 4 months
  Change in RNA in saliva
Immune reponse | 4 months
  Reactions in plasma and saliva will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lynggaard, MD, Principal Investigator — Department of Otolaryngology, Rigshospitalet, University Hospital of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Otolaryngology, Rigshospitalet, University Hospital of Copenhagen, Copenhagen
  - Department of Otolaryngology, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No